CLINICAL TRIAL: NCT00744185
Title: Double Blind, Randomised, Placebo-controlled Study of Propranolol in Infantile Capillary Hemangiomas
Brief Title: Propranolol in Capillary Hemangiomas
Acronym: HEMANGIOMA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely due to some difficulties in recruitment of patients
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2007/27
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Hemangioma, Capillary
Keywords: infantile capillary hemangiomas; propranolol; ultrasonography
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): 30-days placebo treatment
  Interventions: Drug: placebo treatment
- 1 (Experimental): 30-days propranolol treatment
  Interventions: Drug: propranolol treatment

INTERVENTIONS:
Drug: propranolol treatment — 30 days-propranolol treatment : 3 mg/kg 15 days + 4 mg/kg 15 days
  Arms: 1
Drug: placebo treatment — 30 days-placebo treatment : 3 mg/kg 15 days + 4 mg/kg 15 days
  Arms: 2

SUMMARY:
The investigators observed that Propranolol, a beta-blocker commonly used in children was efficient to control the growth of alarming hemangiomas of the face.

The primary objective of this study is to determine the efficiency of 1 month-early treatment of propranolol in infants aged less than 4 months affected by an hemangioma without any consequences on vital or functional structure and not justifying corticosteroids.

The secondary objectives are:

* the kinetic of the hemangioma evolution in infants treated by propranolol
* Observance
* Safety

DETAILED DESCRIPTION:
Infantile hemangiomas are frequent vascular tumors (4 à 10 % of the neonates) and correspond to 100 new cases per year in dermatology consultation of the CHU of Bordeaux. Hemangiomas have a characteristic clinical course marked by early proliferation during 3 to 12 months followed by slow and spontaneous involution from 3 to 7 years. Occasionally, as well as esthetical damages, hemangiomas may impair vital structures, ulcerate, bleed, or cause high-output cardiac failure or significant structural abnormalities. Standard treatments (corticotherapy, interferon, vincristine…) lead to a stagnation of hemangiomas in some cases, but with frequent side effects.

We observed that Propranolol, a beta-blocker usually used in neonates could lead to a decreased in volume of serious haemangiomas of the face (article published in New England Journal of Medicine).

In this study, we proposed to determine the efficiency of 1 month-early treatment of propranolol in neonates aged less than 4 months affected by non alarming hemangioma and not justifying corticotherapy. This is a double blind randomized placebo controlled study of propranolol.

Infants will be recruited from the dermatology consultation of CHU Bordeaux. After verification of eligibility criteria and informed consent of legal surrogates, infants will be randomized to receive either propranolol or either placebo. The infants will be observed during 1 month according to the following visits.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged less than 4 months
* Infant with one or more hemangiomas sized more than 1 cm diameter
* Infant not threatening for vital or functional structure and for which no treatment would be proposed
* Informed consent
* Patient with social insurance.

Exclusion Criteria:

* Alarming hemangioma (s) (complicated forms or localization at risk)
* Cardiac pathology (cardiac malformation, heart failure, cardiac arrhythmias, pulmonary hypertension)
* Asthma
* Bronchopulmonary dysplasia
* Bronchiolitis
* Raynaud syndrome
* Phéochromocytoma
* Development of serious form of hemangioma (bleeding, necrosis, ulceration, infection, respiratory distress) requiring standard treatment

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Proportion of hemangioma thickness variation measured by ultrasonography from the basal state between the two groups after 1 month-treatment. | 30 days treatment

SECONDARY OUTCOMES:
Proportion of hemangioma size variation measured clinically and with photography from the basal state between the two groups after 1 month-treatment. | 30 days-treatment
Observance | 30 days-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Moore, Professor, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Dermatologie Pédiatrique, Bordeaux, France

REFERENCES:
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Background] Tortoriello TA, Snyder CS, Smith EO, Fenrich AL Jr, Friedman RA, Kertesz NJ. Frequency of recurrence among infants with supraventricular tachycardia and comparison of recurrence rates among those with and without preexcitation and among those with and without response to digoxin and/or propranolol therapy. Am J Cardiol. 2003 Nov 1;92(9):1045-9. doi: 10.1016/j.amjcard.2003.06.002. PMID 14583354
- [Background] Villain E, Denjoy I, Lupoglazoff JM, Guicheney P, Hainque B, Lucet V, Bonnet D. Low incidence of cardiac events with beta-blocking therapy in children with long QT syndrome. Eur Heart J. 2004 Aug;25(16):1405-11. doi: 10.1016/j.ehj.2004.06.016. PMID 15321698
- [Background] Kilian K. Hypertension in neonates causes and treatments. J Perinat Neonatal Nurs. 2003 Jan-Mar;17(1):65-74; quiz 75-6. doi: 10.1097/00005237-200301000-00006. PMID 12661740
- [Background] Fritz KI, Bhat AM. Effect of beta-blockade on symptomatic dexamethasone-induced hypertrophic obstructive cardiomyopathy in premature infants: three case reports and literature review. J Perinatol. 1998 Jan-Feb;18(1):38-44. PMID 9527943